CLINICAL TRIAL: NCT04022759
Title: Priming Attachment Security Within an IAPT Setting: A Feasibility and Pilot Study
Brief Title: Priming Attachment Security Within an IAPT Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Charlotte Heathcote, Trainee Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 249633
Record Dates: First submitted 2019-06-17; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Depression
Keywords: Attachment; Improving Access to Psychological Therapies; Security priming
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The feasibility element of the study will aim to explore service users' willingness to participate in the study; clinician's willingness to recruit participants; whether the recruitment method is effective in recruiting participants; and to assess attrition rates.
  The pilot study aims to look at the processes involved in the study as outlined in the protocol, and whether any of these require changes to inform a larger scale RCT; this includes whether the recruitment, randomisation and treatment processes can be carried out effectively. Moreover, the study aims to determine whether the attachment security priming intervention appears to be effective in reducing therapy drop-out; increasing attendance to therapy; and decreasing rates of clients' being stepped-up to step 3 high-intensity services. Secondary to this, the study aims to assess whether priming attachment security appears to have an impact upon levels of depression, anxiety and impaired functioning.
Masking Description: The participant will not explicitly be told which condition they are in by the researcher or the clinician working directly with them. However, they are likely to be able to infer this from the treatment being delivered, having read the information sheet regarding the study. The clinician working with the participant will be aware what condition they are in so that they are able to deliver the appropriate intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Participants randomised to the 'treatment as usual' group will receive behavioural activation guided-self help intervention as routinely delivered in the service.
  Interventions: Behavioral: Treatment as Usual (Behavioural Activation)
- Treatment with Security Prime (Experimental): Participants randomised to the experimental group will receive behavioural activation guided self-help intervention as is routinely delivered in the service with additional attachment security priming intervention.
  Interventions: Behavioral: Treatment as Usual with Security Prime

INTERVENTIONS:
Behavioral: Treatment as Usual with Security Prime — In addition to their treatment as usual (low-intensity guided self-help behavioural activation for depression), participants will complete an initial attachment security priming task during the first session with their allocated clinician. Participants will be prompted in their intervention workbook with a caption regarding what a secure attachment relationship represents. They will be asked to think of a person/ people with whom they feel they have this relationship, and list them. Following this, they are asked to plot these individuals on a diagram of concentric circles in relation to how close they feel this person is to them. The closer to the middle of the diagram the individual places each person, the closer they feel their relationship to that person is.
  Prior to each session with their clinician, they will be prompted to complete a repeated security priming task in order to increase feelings of security prior to therapy sessions.
  Arms: Treatment with Security Prime
Behavioral: Treatment as Usual (Behavioural Activation) — Clients will engage in treatment as usual. This involves low-intensity guided self-help behavioural activation for depression.
  Arms: Treatment as Usual

SUMMARY:
There is growing evidence that priming attachment security is associated with improved attitudes towards therapy, increased engagement and decreased levels of depression and anxiety. Within the Improving Access to Psychological Therapies (IAPT) programme a consistent problem has been identified of high dropout rates at step 2 services (i.e. where mild to moderate anxious and depressed patients receive guided self-help interventions). The current study incorporates a feasibility and pilot design. The feasibility element will explore issues related to study design to determine suitability for conducting a future randomised control trial (RCT). The pilot study will look at the processes outlined in the protocol to determine whether the study components all work together. Moreover, it will preliminarily aim to explore the effectiveness of the attachment security priming intervention on symptoms of depression and anxiety, as well as impaired functioning. Both elements of the study will determine whether any changes are needed to the study design or protocol, and whether a future RCT is suitable and necessary.

DETAILED DESCRIPTION:
The study is being conducted in an IAPT primary care service in North Yorkshire. The study will be recruiting 50 participants experiencing mild to moderate depression who are deemed suitable for 'behavioural activation' low intensity guided self-help intervention. Following telephone screening for intervention, clinicians will ask clients if they wish to hear more about participating in a research study. If participants say yes, their contact details will be passed on to the researcher who will send them the study information sheet and consent form in the post. If the participant consents to taking part in the research, they will be randomised to receive either treatment as usual (low-intensity guided self-help utilising behavioural activation for depression) or treatment with security priming intervention (treatment as usual with an additional security priming task). They will have between 6-8 sessions as routinely delivered within the service and will be asked to complete measures of depression, anxiety and impaired functioning on a sessional basis. The principal investigator at the study site will collect information regarding attendance to therapy, dropout rates, and 'stepping' clients up to higher-intensity therapies as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for Behavioural Activation guided self-help intervention for depression with study NHS IAPT site.
* Over age 18.
* Adequate English ability.

Exclusion Criteria:

* Not suitable for Behavioural Activation guided self-help intervention for depression with study NHS IAPT site.
* Inadequate English ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Attendance | Up to 8 weeks from the beginning to end of treatment
  Number of therapy appointments booked versus number attended for each participant
Dropout | Up to 8 weeks from the beginning to end of treatment
  Number of participants who drop out of therapy after attending at least one session of treatment
Stepping-up to higher intensity services | Up to 8 weeks from the beginning to end of treatment
  The number of participants in the study who are referred for a higher intensity form of therapy during their low-intensity therapy

SECONDARY OUTCOMES:
The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | Weekly for up to 8 weeks from the beginning to end of treatment
  Self-report measure of depression with total possible score ranging from 0 to 27. Scores of 0-4 indicate minimal depression; 5-9 indicates mild depression; 10-14 indicates moderate depression; 15-19 indicates moderately severe depression; and 20-17 indicates severe depression.
The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams, & Lower, 2006) | Weekly for up to 8 weeks from the beginning to end of treatment
  Self-report measure of anxiety with total possible scores between 0 to 21. Scores of 0-5 indicate mild anxiety; 6-10 indicates moderate anxiety; 11-15 indicates moderately severe anxiety; and 16-20 indicates severe anxiety.
The Work and Social Adjustment Scale (WSAS; Mundt, Shear, & Greist, 2002) | Weekly for up to 8 weeks from the beginning to end of treatment
  Self-report measure of impaired functioning with total possible scores of between 0-20. Scores below 10 are associated with subclinical populations. Scores between 10 and 20 indicate significant functional impairment but less severe clinical symptomatology. Scores above 20 indicate moderately severe or worse psychopathology.

CONTACTS AND LOCATIONS:
Overall Officials: James Walton, Principal Investigator — Harrogate IAPT Service
Locations (1):
- Harrogate IAPT Service, Harrogate, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No